CLINICAL TRIAL: NCT03738033
Title: Mobile Education for Emergency Ultrasound
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412004RIND
Record Dates: First submitted 2016-04-27; First posted 2018-11-13 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2018-10

CONDITIONS: Educational Problems
Keywords: emergency medicine ,emergency ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- use of the educational platform: Before the hand-on practice and assessements, the participants use the platform for learning.
  Interventions: Other: educational platform
- without use of the educational platform: Before the hand-on practice and assessements, the participants did not use the platform for learning.

INTERVENTIONS:
Other: educational platform — The platform would be opened before they entered the study.
  Groups: use of the educational platform

SUMMARY:
The investigators aim to investigate the feasibility of using mobile application platform for sonographic education.

Junior physicians at the National Taiwan University Hospital will be enrolled in this study. To design and develop a secure mobile application platform (consisting of mobile device and a cloud-based server) for interactive teaching, remote social-based consultation and discussion. The information exchange through the platform carries images and simulated cases.

This pioneer study can provide experience of mobile sonographic education and contribute to current medical education. Moreover, it can improve decision-making process and quality of care, and could lessen crowdedness at emergency departments. Furthermore, the integrated platform can be used in other educational programs in the future.

DETAILED DESCRIPTION:
As usual, it takes time for junior emergency physicians to have good diagnostic accuracy through traditional sonographic education. Applying the technology built in this project, junior emergency physicians will be provided with intelligent learning programs anywhere and anytime.

Junior physicians at the National Taiwan University Hospital will be enrolled in this study.

ELIGIBILITY:
Inclusion criteria:

The junior physicians of the department of emergency medicine of the National Taiwan University Hospital.

Exclusion criteria:

The junior physicians of the department of emergency medicine of the National Taiwan University Hospital, refused to enter the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The junior physicians of the department of emergency medicine of the National Taiwan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
assessment for ultrasound scanning | one week
  use 5-point Likert scale (1 to 5 scores)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Che Wu, Dr, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lien WC, Lin P, Chang CH, Wu MC, Wu CY. The effect of e-learning on point-of-care ultrasound education in novices. Med Educ Online. 2023 Dec;28(1):2152522. doi: 10.1080/10872981.2022.2152522. PMID 36433837